CLINICAL TRIAL: NCT02899208
Title: Can an Actigraph be Used to Predict Physical Function in Intensive Care Patients?
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SE 3-16
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Critical Illness; Quality of Life; Physical Activity
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to investigate whether an actigraph, measuring in-hospital activity, used for a week after discharge from the ICU at Zealand University Hospital Køge, can predict physical function at three-month follow up.

The hospital activity will be measured with actigraphy, a measurement tool that quantifies activity level. The activity will be measured for 7 days after ICU discharge. The actigraph is to be worn as a bracelet.

The physical function will be measured with Chelsea Critical Care Physical Assessment Tool (CPAx). CPAx is assessed at ICU discharge and after three months.

DETAILED DESCRIPTION:
Treatment at an Intensive Care Unit (ICU) is often needed for the survival of critically ill patients, but it can take a long time to recover. A number of high quality studies have shown that patients experience functional impairments for a long period after discharge, even for years.

These patients may suffer from a number of other negative influences of their critical illness and ICU stay, e.g. memory problems, episodes of depression, cognitive dysfunction and sleeping disorders. These symptoms are seen in both medical and surgical patients and has been named the Post Intensive Care Syndrome.

Physical rehabilitation is important and must start already during admission, in order to regain some of the function and independence of the patients. This has a well documented effect on both mental and physical wellbeing.

Actigraphy is a newer way of quantifying the activity level continuously. It is validated and has been used in the ICU to assess agitation and sedation and in an oncological, surgical and even an ICU population to assess sleep.

It is easy to use, non-invasive and inexpensive. It is worn like a bracelet and doesn't impair the patients mobility or ambulation.

Another issue when evaluating physical impairments is the choice of method for assessing physical function. For this study, the investigators use the Chelsea Critical Care Physical Assessment Tool (CPAx) as it has good validity and clinimetric properties and is easy to use. Also, it can be done as part of the daily training as it is developed specifically for the ICU.

The aim of this study is to investigate how the in-hospital activity level of patients after ICU discharge is associated with their physical function at three months post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Admitted to the ICU for > 24 h

Exclusion Criteria:

* Not able to speak and understand Danish
* Patients suffering from dementia or psychosis
* Discharged from the ICU to terminal care
* Patients transferred to another hospital during ICU stay
* Patients living outside the Region of Zealand
* Patients suffering from total paralysis before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU at Zealand University Hospital, Køge, in the study period
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
The association between actigraph levels and CPAx at three months after discharge from ICU | 3 months after discharge from intensive care unit
  The association between actigraph levels and CPAx score (from 0 to 50 points)

SECONDARY OUTCOMES:
CPAx at discharge from ICU | Within 24 hours of discharge from intensive care unit
  CPAx score (from 0 to 50 points)
Activity measured with actigraph during one week after ICU-discharge | One week after discharge from ICU
  Activity measured with an actigraph watch placed on the patients' wrist
Association between early activity level measured with actigraphy for 7 days and SF 36 at three months after discharge from ICU | 3 months after discharge from intensive care unit
  The association between actigraph levels and SF-36 score
Association between early activity level measured with actigraphy for 7 days and Hospital Anxiety and Depression Scale (HADS) at three months after discharge from ICU | 3 months after discharge from intensive care unit
  The association between actigraph levels and HADS score (from 0 to 42 points)
Association between early activity level measured with actigraphy for 7 days and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) at three months after discharge from ICU | 3 months after discharge from intensive care unit
  The association between actigraph levels and RBANS score
Association between early activity level measured with actigraphy for 7 days and mortality within hospital stay, after ICU discharge | The period within hospital stay, after intensive care unit discharge
  The association between actigraph levels and hospital mortality
Association between early activity level measured with actigraphy for 7 days and mortality within 90 days after ICU discharge | 3 months after discharge from intensive care unit
  The association between actigraph levels and 90-day mortality
Association between early activity level measured with actigraphy for 7 days and consumption of opioids (strong/weak) at 90 days follow up. | 3 months after discharge from intensive care unit
  The association between actigraph levels and opioid-consumtion (morphine-equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: Stine Estrup, MD, Principal Investigator — Zealand University Hospital, Køge Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Grap MJ, Borchers CT, Munro CL, Elswick RK Jr, Sessler CN. Actigraphy in the critically ill: correlation with activity, agitation, and sedation. Am J Crit Care. 2005 Jan;14(1):52-60. PMID 15608109
- [Background] Parry SM, Granger CL, Berney S, Jones J, Beach L, El-Ansary D, Koopman R, Denehy L. Assessment of impairment and activity limitations in the critically ill: a systematic review of measurement instruments and their clinimetric properties. Intensive Care Med. 2015 May;41(5):744-62. doi: 10.1007/s00134-015-3672-x. Epub 2015 Feb 5. PMID 25652888
- [Background] Corner EJ, Wood H, Englebretsen C, Thomas A, Grant RL, Nikoletou D, Soni N. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013 Mar;99(1):33-41. doi: 10.1016/j.physio.2012.01.003. Epub 2012 Mar 30. PMID 23219649
- [Background] Corner EJ, Soni N, Handy JM, Brett SJ. Construct validity of the Chelsea critical care physical assessment tool: an observational study of recovery from critical illness. Crit Care. 2014 Mar 27;18(2):R55. doi: 10.1186/cc13801. PMID 24669784
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092